CLINICAL TRIAL: NCT04354207
Title: Comparative Study of Vitamin D and Its Receptor Gene Polymorphisms in Lithuanian, Latvian, and Taiwanese Children and Adults With Atopic Dermatitis and Asthma
Brief Title: Vitamin D and Its Receptor Gene Polymorphisms in Lithuanian, Latvian and Taiwanese Patients With Atopic Dermatitis and Asthma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Research Council of Lithuania (Other)
Responsible Party: Principal Investigator, Brigita Sitkauskiene, Prof., Head of Department of Immunology and Allergology, Lithuanian University of Health Sciences
Other Study IDs: LLTADA; S-LLT-20-1 (Other Grant/Funding Number: Researh Council of Lithuania)
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Atopic Dermatitis; Asthma
MeSH Terms: conditions — Dermatitis, Atopic; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Atopic dermatitis
  Interventions: Diagnostic Test: Peripheral vein punction; Diagnostic Test: Stool collection
- Asthma
  Interventions: Diagnostic Test: Peripheral vein punction; Diagnostic Test: Stool collection
- Healthy individuals
  Interventions: Diagnostic Test: Peripheral vein punction; Diagnostic Test: Stool collection

INTERVENTIONS:
Diagnostic Test: Peripheral vein punction — Vitamin D level, vitamin D receptor genetic polymorphisms, allergen specific IgE and total IgE will be measured in peripheral blood
Diagnostic Test: Stool collection — Gut microbiome will be investigated in stool samples.

SUMMARY:
The role of vitamin D is well known in calcium and phosphate homeostasis; however, in addition to traditional functions, vitamin D has an important role in pathogenesis of different allergic diseases, such as asthma, atopic dermatitis (AD), and food allergy. There are evidences that lower cord blood vitamin D status is observed in infants with eczema. More-over, vitamin D level is decreased in subjects with asthma. One of the most important functions of vitamin D is to modulate the immune system response, both innate and adaptive, by suppressing Th2-type response and increasing natural killer cells. Vitamin D induces a higher level of IL-10, which is known as anti-inflammatory cytokine. Other studies have shown that vitamin D contributes to the conversion of CD4+ T cells to T regulatory cells. Recent studies showed that higher serum 25-hydroxyvitamin D level was associated with a reduced risk of asthma exacerbation and hospitalization. Vitamin D can enhance dexamethasone-induced MAP kinase phosphatase-1 (MKP-1) expression in peripheral blood mononuclear cells. Experimental data suggest that vitamin D can potentially increase the therapeutic response to glucocorticoid and can be used as an add-on treatment in steroid-resistant asthmatics. Vitamin D stimulates the production and regulation of skin antimicrobial peptides, such as cathelicidins, which have both direct antimicrobial activity and induced host cellular response by triggering cytokine release. Recent evidence suggests that low blood vitamin D level is a risk factor for food allergy.

Vitamin D acts by binding to the vitamin D receptors (VDRs), which are located in a variety of tissues. VDRs have been identified on nearly all cells of the immune system including T cells, B cells, neutrophils, macrophages, and dendritic cells (DCs).

Vitamin D deficiency predisposes to gastrointestinal infections by changing gut micro-biota, which may promote the development of food allergy. However the detail mechanism how vitamin D affects or protects the development of allergic diseases is still unknown. Vitamin D level is determined by sun exposure.

Due to the fact that Lithuania, Latvia and Taiwan are located in different latitudes of north hemisphere with markedly different sun exposure, in this Joint collaboration study between Taiwan, Lithuanian and Latvia, we are going to study, (1). Serum vitamin D level in children and adults with AD and/or asthma in Lithuania, Latvia and Taiwan. (2). VDRs genetic polymorphisms of AD and/or asthma in children and adults in Lithuania, Latvia and Taiwan. (3). Finally, we would like to explore the gut microbiome of patients with AD and/or asthma in Lithuanian, Latvian and Taiwanese children and adults; and to estimate possible relationship between gut microbiome and vitamin D level and VDRs genetic polymorphisms. We believe that this study will be the first which compares the populations with different geographical and ecological factors having the same allergic diseases. We hope that these results will provide the answer about the role of vitamin D in the prevention, or in the future, in treatment of allergic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate asthma
* Patients with mild to moderate atopic dermatitis
* Healthy individuals

Exclusion Criteria:

* Acute or chronic infections
* Oncological diseases
* Acute systemic autoimmune diseases
* Use of systemic immunosuppressants (wait 1 month)
* Use of vitamin D supplementation
* Use of systemic antihistamines (wait 1 week)

Max Age: 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adults with mild to moderate asthma or mild to moderate atopic dermatits.
  Healthy individuals as control group.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin D level in serum in patients with atopic dermatitis, asthma and healthy individuals from Lithuania, Latvia and Taiwan | 2nd year of study
  Comparison of serum vitamin D level (25(OH)D) by ELISA between studied groups
Vitamin D receptors (VDRs) genetic polymorphisms in patients with atopic dermatitis, asthma and healthy individuals from Lithuania, Latvia and Taiwan | 2nd year of study
  Comparison of VDRs genetic polymorphisms using genetic evaluation between studied groups
Composition of gut microbiome in patients with atopic dermatitis, asthma and healthy individuals from Lithuania, Latvia and Taiwan | 3rd year of study
  Investigation and comparison of gut microbiome using genetic evaluation between studied groups

CONTACTS AND LOCATIONS:
Overall Officials: Brigita Sitkauskiene, Prof., Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No